CLINICAL TRIAL: NCT04924608
Title: A Phase III, Multicentre, International Study With a Parallel, Randomised, Double-blind, Placebo-controlled, 2 Arm Design to Assess the Efficacy and Safety of Selumetinib in Adult Participants With NF1 Who Have Symptomatic, Inoperable Plexiform Neurofibromas (KOMET)
Brief Title: Efficacy and Safety of Selumetinib in Adults With NF1 Who Have Symptomatic, Inoperable Plexiform Neurofibromas
Acronym: KOMET
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D134BC00001; 2020-005607-39 (EudraCT Number)
Record Dates: First submitted 2021-05-14; First posted 2021-06-14 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Neurofibromatosis 1; Plexiform Neurofibroma (PN)
Keywords: Neurofibromatosis Type 1; NF1; Plexiform Neurofibroma (PN); PNs; Selumetinib; MEK inhibitor
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform | interventions — AZD 6244

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Selumetinib
  Interventions: Drug: Selumetinib
- Arm B (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Selumetinib — Selumetinib oral capsules (10 mg and 25 mg)
  Other Names: AZD6244
  Arms: Arm A
Other: Placebo — Placebo oral capsules for Selumetinib masking (10 mg and 25 mg)
  Arms: Arm B

SUMMARY:
A global study to demonstrate the effectiveness of selumetinib in participants with NF1 who have symptomatic, inoperable plexiform neurofibromas.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, 2 arm multicentre, global Phase III study to assess the efficacy and safety of selumetinib compared with placebo in adult participants with NF1 who have symptomatic, inoperable PN.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults ≥ 18 years at enrollment with diagnosis of NF1 with symptomatic, inoperable PN
* At least one inoperable target PN measurable by volumetric MRI analysis
* Chronic target PN pain score documented for minimum period during screening period
* Stable chronic PN pain medication use at enrollment
* Adequate organ and marrow function

Key Exclusion Criteria:

* Confirmed or suspected malignant glioma or MPNST (low grade glioma, including optic glioma not requiring systemic therapy or radiation therapy are exempt from this exclusion)
* History of malignancy except for malignancy treated with curative intent with no known active disease ≥ 5 years before the first dose of study intervention and of low potential risk for recurrence
* Clinically significant cardiovascular disease, including inherited coronary disease, acute coronary syndrome within 6 months prior to enrollment, uncontrolled angina, symptomatic heart failure, cardiomyopathy, severe valvular heart disease, abnormal LVEF and uncontrolled hypertension
* Ophthalmological findings/conditions including intraocular pressure > 21 mmHg, RPED/CSR or RVO
* Prior exposure to MEK inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2029-02-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alice P. Chen, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (32):
- United States (4):
  - Research Site, Gainesville, Florida
  - Research Site, Rockville, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Commack, New York
- Australia (2):
  - Research Site, Melbourne
  - Research Site, St Leonards
- Brazil (3):
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São Paulo
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (3):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Shenyang
- France (3):
  - Research Site, Créteil
  - Research Site, Lyon
  - Research Site, Toulouse
- Germany (3):
  - Research Site, Hamburg
  - Research Site, Tübingen
  - Research Site, Würzburg
- Italy (3):
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
- Japan (3):
  - Research Site, Minatoku
  - Research Site, Nagoya
  - Research Site, Shinjuku-ku
- Research Site, Bydgoszcz, Poland
- Research Site, Moscow, Russia
- Spain (2):
  - Research Site, Badalona
  - Research Site, Madrid
- United Kingdom (2):
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Chen AP, Coyne GO, Wolters PL, Martin S, Farschtschi S, Blanco I, Chen Z, Darrigo LG Jr, Eoli M, Whittle JR, Nishida Y, Lamarca R, de la Rosa Rodriguez R, Adeyemi A, Herrero I, Llorente N, Diede SJ, Dombi E, Wolkenstein P; KOMET study investigators. Efficacy and safety of selumetinib in adults with neurofibromatosis type 1 and symptomatic, inoperable plexiform neurofibromas (KOMET): a multicentre, international, randomised, placebo-controlled, parallel, double-blind, phase 3 study. Lancet. 2025 Jun 21;405(10496):2217-2230. doi: 10.1016/S0140-6736(25)00986-9. Epub 2025 Jun 2. PMID 40473450
- See also: Redacted Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D134BC00001&attachmentIdentifier=e31a38ab-227e-4a34-8fce-3cc35a30caa4&fileName=D134BC00001_-_KOMET-Clinical_Study__Protocol-v.4__Redacted-updated-30Jul25-PDF-A.pdf&versionIdentifier=
- See also: Redacted Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D134BC00001&attachmentIdentifier=40eea1cc-cd65-427a-8134-01b9f22fa5c2&fileName=D134BC00001_-___Statistical_Analysis_Plan_Redacted-PDF-A.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D134BC00001&attachmentIdentifier=352b6ecb-e92a-42fe-9449-794475579d93&fileName=D134BC00001_(KOMET)_Primary_Analysis_CSR_Synopsis-30Jul25_Redacted-PDF-A.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Selumetinib 25 mg/m2; Placebo: Actual Treatment Group
Period: Overall Study
Arm/Group | Selumetinib 25 mg/m2 | Placebo
Started | 71 | 74
Completed | 0 | 0
Not Completed | 71 | 74
Not completed — Adverse Event | 10 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Ongoing at the data cut-off date | 54 | 60
Not completed — Progressive Disease | 2 | 0
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Other reason | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selumetinib 25 mg/m2 | Placebo | Total
Number analyzed (Participants) | 71 | 74 | 145
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were collected at screening period
  Years | 32.6 (11.42) | 29.8 (8.72) | 31.2 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics were collected at screening period
  Participants
    Female | 38 | 32 | 70
    Male | 33 | 42 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Baseline characteristic were collected at screening period
  Participants
    Hispanic or Latino | 5 | 9 | 14
    Not Hispanic or Latino | 63 | 63 | 126
    Unknown or Not Reported | 3 | 2 | 5
Baseline PAINS-pNF chronic target PN pain intensity score [Number; unit: Participants] — The PAINS-pNF (Pain Intensity Scale for Plexiform Neurofibroma) chronic target PN pain intensity measures the participants' experience of chronic PN-related pain intensity with score from 0 (no chronic tumor pain) to 10 (worst chronic tumor pain). Baseline characteristics were collected at screening period.
  Participants
    Baseline PAINS-pNF chronic target PN pain intensity score >= 3 | 50 | 53 | 103
    Baseline PAINS-pNF chronic target PN pain intensity score < 3 | 21 | 21 | 42
Height [Mean (Standard Deviation); unit: cm] — Baseline characteristics were collected at screening period
  cm | 163.517 (9.3702) | 165.798 (12.2517) | 164.698 (10.9784)
Weight [Mean (Standard Deviation); unit: kg] — Baseline characteristics were collected at screening period
  kg | 65.896 (15.9763) | 66.271 (17.3971) | 66.087 (16.6596)
BSA [Mean (Standard Deviation); unit: m^2] — Baseline Body Surface Area. Baseline characteristics were collected at screening period
  m^2 | 1.713 (0.2319) | 1.732 (0.2620) | 1.722 (0.2471)
Geographical region [Number; unit: count] — Baseline characteristics were collected at screening period
  count
    China | 11 | 13 | 24
    Europe (includes France, Germany, Italy, Poland, Russia, Spain, and United Kingdom) | 31 | 30 | 61
    Japan | 7 | 8 | 15
    Rest of World (includes Australia, Brazil, Canada, and United States) | 22 | 23 | 45
Race [Number; unit: Participants] — Baseline characteristics were collected at screening period
  Participants
    Asian | 22 | 23 | 45
    Black or African American | 6 | 3 | 9
    White | 38 | 43 | 81
    Other | 2 | 3 | 5
    Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Partial and Complete Response Rate (ORR) by End of Cycle 16 Using Volumetric MRI Analysis as Determined by ICR (Per REiNS Criteria) in Participants With NF1 Who Have Symptomatic, Inoperable PN.
Description: Objective response rate is defined as the proportion of participants who have a confirmed CR (defined as disappearance of the target PN, confirmed by a consecutive scan within 3 to 6 months after the first response) or confirmed PR (defined as a target PN volume decrease ≥ 20%, compared to baseline, confirmed by a consecutive scan within 3 to 6 months after the first response) by end of Cycle 16 as determined by ICR per REiNS criteria.
  Increase in the volume of the target PN by 20% or more compared to baseline or the time of best response after documenting a PR is considered as PD.
Time Frame: From first dose up until progression (if it occurs prior to the end of Cycle 16), or the last evaluable assessment up to and including the end of Cycle 16, excluding MRI during prolonged study intervention interruption (defined as interruption >= 28 days)
Population: Full analysis set - All patients who are randomized to study intervention
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Selumetinib 25 mg/m2 | Placebo
Number analyzed (Participants) | 71 | 74
Percentage | 19.7 [11.2 to 30.9] | 5.4 [1.5 to 13.3]
Statistical Analysis 1: Comparison: Selumetinib 25 mg/m2 vs Placebo; Test type: Superiority; p = 0.0112, Fisher Exact; The ORR will be compared at the end of Cycle 16 between selumetinib vs placebo with the 2-sided significance level 0.047

2. Secondary Outcome: (First Key Secondary) The Difference of the Means in the Change From Baseline in PAINS-pNF Chronic Target PN Pain Intensity Score at Cycle 12 Between Selumetinib and Placebo, Primary Analysis
Description: The PAINS-pNF (Pain Intensity Scale for Plexiform Neurofibroma) chronic target PN pain intensity measures the participants' experience of chronic PN-related pain intensity with score from 0 (no chronic tumor pain) to 10 (worst chronic tumor pain). Baseline PAINS-pNF chronic target PN pain score is defined as the average of the available daily PAINS-pNF chronic target PN pain scores in the screening perio, while for Cycle 12, it is defined as the average of the available daily scores for the 28-days cycle up to and including the last day assessment of cycle 12. The difference of the means in the change from baseline at Cycle 12 between selumetinib and placebo in participants with a PAINS-pNF chronic target PN pain score of ≥ 3 at baseline is presented.
Time Frame: Baseline and end of cycle 12 of study intervention
Population: Pain full analysis set - subjects randomised to study intervention with a baseline PAINS-pNF chronic target PN pain intensity score >= 3.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Selumetinib 25 mg/m2 | Placebo
Number analyzed (Participants) | 42 | 42
Scores on a scale | -2.0 (0.30) | -1.3 (0.29)
Statistical Analysis 1: Comparison: Selumetinib 25 mg/m2 vs Placebo; Test type: Superiority; p = 0.070, Mixed Models Analysis; Analysis is based on a MMRM model for repeated measures, Kenward-Roger method is used to estimate the degrees of freedom; LS mean difference = -0.8, 95% CI 2-sided [-1.6 to 0.1], Standard Error of Mean 0.41

3. Secondary Outcome: (First Key Secondary) The Difference of the Means in the Change From Baseline in PAINS-pNF Chronic Target PN Pain Intensity Score at Cycle 12 Between Selumetinib and Placebo, Supplemental Analysis
Description: The PAINS-pNF (Pain Intensity Scale for Plexiform Neurofibroma) chronic target PN pain intensity measures the participants' experience of chronic PN-related pain intensity with score from 0 (no chronic tumor pain) to 10 (worst chronic tumor pain). Baseline PAINS-pNF chronic target PN pain score is defined as the average of the available daily PAINS-pNF chronic target PN pain scores in the screening perio, while for Cycle 12, it is defined as the average of the available daily scores for the 28-days cycle up to and including the last day assessment of cycle 12. The difference of the means in the change from baseline at Cycle 12 between selumetinib and placebo participants is presented.
Time Frame: Baseline and end of cycle 12 of study intervention
Population: Full analysis set - subjects randomised to study intervention
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Selumetinib 25 mg/m2 | Placebo
Number analyzed (Participants) | 57 | 62
Scores on a scale | -1.6 (0.22) | -0.9 (0.21)
Statistical Analysis 1: Comparison: Selumetinib 25 mg/m2 vs Placebo; supplementary analysis is not controlled for multiplicity; Test type: Superiority; p = 0.024, Mixed Models Analysis — nominal; [statistical method as in outcome 2, analysis 1]; LS mean difference = -0.7, 95% CI 2-sided [-1.3 to -0.1], Standard Error of Mean 0.30

4. Secondary Outcome: (Second Key Secondary Endpoint) The Difference of the Means in the Change From Baseline in PlexiQoL Total Score at Cycle 12
Description: PlexiQoL (Plexiform Neurofibroma Quality of Life scale) is a patient-derived QoL measure specific to adults with NF1-associated PNs. It assesses the impact of PNs on patients' ability to fulfil their human needs. The measure consists of 18 dichotomous items with 0 =Not True and 1 = True. PlexiQoL total scores were calculated by the sum of all items to a maximum of 18, with lower scores indicating better quality of life. The change from baseline to the end of each cycle in PlexiQoL total score was derived as the PlexiQoL total score at the cycle 12 minus baseline PlexiQoL total score and presented.
Time Frame: Baseline and end of Cycle 12 of study intervention
Population: Full analysis set - subjects randomised to study intervention
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Selumetinib 25 mg/m2 | Placebo
Number analyzed (Participants) | 57 | 59
Scores on a scale | -0.4 (0.45) | -0.3 (0.44)
Statistical Analysis 1: Comparison: Selumetinib 25 mg/m2 vs Placebo; Test type: Superiority; p = 0.918, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; LS mean difference = -0.1, 95% CI 2-sided [-1.2 to 1.1], Standard Error of Mean 0.59

ADVERSE EVENTS:
Time Frame: All-cause mortality (death due to any cause) and Treatment emergent adverse events during randomised period, which is from the first dose of study intervention until the first date when selumetinib kit(s) are dispensed at Cycle 12 Day 28 (about 1 year), or 30 days after study intervention discontinuation, or up to one day prior to start of subsequent therapy, whichever occurs first. The medians of total treatment duration were 336 days for Selumetinib group and 335 days for Placebo group.
Description: All-cause mortality was reported for all subjects. Adverse events were reported for subjects who received at least one dose of study drug and include AEs that start prior to and worsen after treatment or with an onset or worsening date on or after the date of first selumetinib dose up to and including 30 days after the date of last selumetinib dose. All TESAE, and non-serious TEAEs for a preferred term at a frequency of > 5% in any treatment group during the randomized period are presented.
Arm/Group | Selumetinib 25 mg/m2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/74
Serious Adverse Events (participants affected / at risk) | 10/71 | 9/74
Other Adverse Events (participants affected / at risk) | 70/71 | 54/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selumetinib 25 mg/m2 (N=71) | Placebo (N=74)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neurofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Neurofibrosarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selumetinib 25 mg/m2 (N=71) | Placebo (N=74)
Vomiting (Gastrointestinal disorders) | 18 (33) | 6 (7)
Fatigue (General disorders) | 14 (14) | 10 (10)
Oedema peripheral (General disorders) | 11 (14) | 1 (1)
Pyrexia (General disorders) | 5 (6) | 3 (3)
Covid-19 (Infections and infestations) | 11 (12) | 15 (16)
Paronychia (Infections and infestations) | 9 (9) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 5 (6)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 8 (10)
Alanine aminotransferase increased (Investigations) | 11 (12) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 13 (17) | 4 (5)
Blood creatine phosphokinase increased (Investigations) | 32 (40) | 4 (6)
Ejection fraction decreased (Investigations) | 5 (5) | 2 (3)
Protein urine present (Investigations) | 0 (0) | 4 (5)
Weight increased (Investigations) | 4 (4) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 6 (8) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (9)
Headache (Nervous system disorders) | 7 (8) | 9 (18)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (7) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (14) | 8 (8)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 42 (49) | 8 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 13 (15) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (7)
Rash (Skin and subcutaneous tissue disorders) | 11 (16) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 30 (50) | 9 (9)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 18 (19) | 12 (14)
Stomatitis (Gastrointestinal disorders) | 7 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-11-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT04924608/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT04924608/SAP_001.pdf